CLINICAL TRIAL: NCT07309913
Title: China Atrial Fibrillation With Complex Metabolic Disorders Cohort Study (CAME Cohort)
Brief Title: China Atrial Fibrillation With Complex Metabolic Disorder Cohort Study (CAME Cohort)
Acronym: CAME Cohort
Status: Not yet recruiting | Type: Observational
Sponsor: Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Other Study IDs: 2025101847
Record Dates: First submitted 2025-11-23; First posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-11

CONDITIONS: Atrial Fibrillation (AF); Metabolic Disorders
MeSH Terms: conditions — Atrial Fibrillation; Metabolic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples Without DNA — peripheral blood
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- No metabolic disorder
- Single metabolic disorder
- Complex metabolic disorder (≥2 types)

SUMMARY:
The number of atrial fibrillation (AF) patients in China is approximately 32.76 million, with a prevalence rate of 2.3%. AF is associated with severe outcomes such as stroke and heart failure. Metabolic disorders (e.g., obesity, diabetes mellitus, dyslipidemia) are closely linked to the onset and prognosis of AF. However, the epidemiological characteristics and disease burden of AF combined with metabolic disorders in China remain unclear. Additionally, the impact of complex multi-dimensional metabolic disorders on AF prognosis requires further investigation, and current clinical guidelines lack targeted management recommendations for this population.

ELIGIBILITY:
Inclusion Criteria

* Meet the diagnostic criteria for atrial fibrillation: Single-lead electrocardiogram (≥30 seconds) or 12-lead electrocardiogram (≥10 seconds) shows disappearance of P waves, replaced by fibrillation waves (f waves) with irregular amplitude, morphology and duration, and absolutely irregular RR intervals.
* Aged ≥ 18 years.
* Willing to sign the informed consent form and cooperate with long-term follow-up.

Exclusion Criteria

* Suffering from infective endocarditis or myocarditis.
* Having clear etiological factors of atrial fibrillation caused by hyperthyroidism, and the etiology has not been effectively controlled.
* Suffering from severe mental illness and being unable to comply with the study requirements.
* Pregnant women.
* Patients with malignant tumors or substance abuse (e.g., cocaine, heroin).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Meets the diagnostic criteria for AF: single-lead electrocardiogram (ECG) ≥ 30 seconds or 12-lead ECG ≥ 10 seconds, with disappearance of P waves, presence of fibrillatory (f) waves, and absolute irregularity of RR intervals.
Sampling Method: Probability Sample
Enrollment: 3459 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2036-02-01 (Estimated); Study Completion 2036-06-01 (Estimated)

PRIMARY OUTCOMES:
Major Adverse Cardiovascular Events (MACE) | From enrollment to the end of follow-up at 5 years
  Major Adverse Cardiovascular Events (MACE) - Composite outcome including the following components, all assessed during the entire follow-up period:
  * All-cause mortality: Defined as any death regardless of cause, confirmed by death certificate, medical records or family report.
  * Stroke: Defined as acute focal neurological deficit lasting ≥24 hours (or leading to death within 24 hours) due to cerebral infarction or intracerebral hemorrhage, confirmed by cranial computed tomography (CT) or magnetic resonance imaging (MRI).
  * Heart failure-related hospitalization: Defined as hospitalization requiring inpatient treatment due to worsening heart failure symptoms (e.g., dyspnea, edema), with objective evidence of heart failure exacerbation (e.g., elevated BNP, pulmonary congestion on chest imaging).

SECONDARY OUTCOMES:
Cardiovascular mortality | From enrollment to the end of follow-up at 5 years
  Defined as death caused by cardiovascular diseases (including myocardial infarction, heart failure, stroke, arrhythmia, etc.), determined by review of death certificate, autopsy report or clinical records by the endpoint adjudication committee.
Cognitive impairment assessed by the Mini-Mental State Examination (MMSE) scale | From enrollment to the end of follow-up at 5 years
  Defined as a score ≤23 on the Mini-Mental State Examination (MMSE) scale at follow-up visits, with cognitive decline confirmed by a neuropsychological assessment panel if necessary (MMSE covers orientation, memory, attention, calculation, language and motor functions).
Quality of life: Assessed by the Atrial Fibrillation Effect on Quality of Life (AFEQT) questionnaire | From enrollment to the end of follow-up at 5 years
  Assessed by the Atrial Fibrillation Effect on Quality of Life (AFEQT) questionnaire at baseline, 6 months, 12 months and annually thereafter; total score ranges from 0 (worst quality of life) to 100 (best quality of life), with subscores for symptoms, activity, treatment concern and quality of life reported separately.
Atrial fibrillation (AF) treated with catheter ablation for 2 or more times | From enrollment to the end of follow-up at 5 years
  Defined as receiving a second or subsequent catheter ablation procedure due to AF recurrence after the initial ablation, documented by interventional procedure records.